CLINICAL TRIAL: NCT06097637
Title: Underwater Endoscopic Mucosal Resection Versus Metal Clips With Hot Snare Polypectomy for Resection of Big Pedunculated Colorectal Polyps: A Randomized Controlled Trial
Brief Title: Underwater Endoscopic Mucosal Resection Versus Metal Clips With Hot Snare Polypectomy for Resection of Big Pedunculated Colorectal Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-139A-YJ01
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-07

CONDITIONS: Pedunculated Colorectal Polyps; Haemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- underwater endoscopic mucosal resection (Experimental): underwater endoscopic mucosal resection for resection of big pedunculated colorectal polyps
  Interventions: Other: underwater endoscopic mucosal resection
- hot snare polypectomy (Active Comparator): hot snare polypectomy for resection of big pedunculated colorectal polyps
  Interventions: Other: hot snare polypectomy

INTERVENTIONS:
Other: underwater endoscopic mucosal resection — underwater endoscopic mucosal resection achieves similar rates of complete resection with comparable safety, with lower rates of recurrence and fewer repeat procedures.
  Arms: underwater endoscopic mucosal resection
Other: hot snare polypectomy — Current guidelines recommend preoperative hot snare polypectomy after preoperative saline injection, nylon ring, or metal clip ligation of the tip and pedicle of the polyps
  Arms: hot snare polypectomy

SUMMARY:
Endoscopic resection of pedunculated polyps mainly focuses on how to prevent bleeding, and also needs to pay attention to the convenience of resection and the integrity of resection, which means that different endoscopic resection strategies should be adopted for pedunculated polyps with different pedicle sizes. The head larger than 20mm or pedicle larger than 5mm are defined as large pedunculated polyps, which are at greater risk of bleeding. Current guidelines recommend hot removal by snare following preoperative saline injection, ligation of the pedicle with a nylon ring or metal clip, depending on the size of the polyp head and pedicle. However, the use of snares and metal clamps does not appear to reduce delayed postoperative bleeding, and the technical requirements of nylon ligation are relatively high. Recent studies have found that Underwater endoscopic mucosal resection (UEMR) is also safe and effective for the treatment of large and medium colorectal sessile polyps. Therefore, it is still necessary to further explore new safe and effective endoscopic resection strategies and techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing endoscopic resection of small and medium pedicled polyps in the First Affiliated Hospital of Ningbo University from October 2023 to August 2026;
2. Age 18-75 years old;
3. Patients who voluntarily agreed to participate in this study and signed informed consent.

Exclusion Criteria:

1. Persons under 18 years of age
2. Persons unwilling or unable to provide informed consent
3. Treatment or radiotherapy for malignant diseases, severe chronic heart or lung diseases, coronary or cerebrovascular events requiring hospitalization within the last 3 months
4. Malignant polyps have infiltrated the pedicle
5. Abdominal symptoms such as severe abdominal pain, abdominal distension, and nausea
6. Patients with inadequate intestinal preparation
7. Patients with lifelong anticoagulant therapy or severe bleeding diseases, patients who have recently taken anticoagulant drugs or antiplatelet drugs (within 1 week)
8. Pregnant or lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of immediate bleeding | 1 Minutes
  Immediate bleeding was defined as an intraoperative bleeding immediately after Immediate bleeding staging: If there is no bleeding, fill in 'none'; Level 1, spontaneous hemostasis within 60 seconds; Level 2, continuous small bleeding for more than 60 seconds; Level 3, continuous bleeding for more than 60 seconds requires endoscopic treatment; Level 4, arterial spray

SECONDARY OUTCOMES:
delayed hemorrhage | 2 weeks and 4 weeks
  Any symptoms of gastrointestinal bleeding (e. g. hematochezia) occurred within 30 days after polypectomy and were classified as mild or severe according on the severity of the bleeding

OTHER OUTCOMES:
Immediate perforation rate | 30 seconds
  perforation

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China